CLINICAL TRIAL: NCT02055144
Title: An Exploratory Study of the Performance of Mass-Spectrometry Based Test Veristrat in Prediction of Benefit of First Line NSCLC Patients From Treatment With Standard Chemotherapy Regimens
Brief Title: Veristrat as Predictor of Benefit of First Line Non Small Cell Lung Cancer (NSCLC) Patients From Standard Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy (Other)
Responsible Party: Principal Investigator, Francesco Grossi, MD, IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Other Study IDs: VERISTRAT/IST
Record Dates: First submitted 2014-01-30; First posted 2014-02-04 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Non Small Cell Lung Cancer
Keywords: NSCLC; VeriStrat; chemotherapy; circulating tumor cells
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplastic Cells, Circulating

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples, urine samples, circulating tumour cells from peripheral blood. Such samples will be obtained before start of treatment (within 2 weeks), and at each patient's evaluation and at progression
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non squamous histology: patients with advanced, non-squamous non-small cell lung cancer treated with cisplatin (or carboplatin) and pemetrexed. Maintenance with pemetrexed is allowed.
- Squamous histology: patients with advanced squamous non-small cell lung cancer treated with cisplatin (or carboplatin) and gemcitabine

SUMMARY:
VeriStrat® is a pretreatment blood-based test correlated with clinical outcome after EGFR-TKI therapy in non-small cell lung cancer (NSCLC) patients.

The investigators hypothesis is that VeriStrat could be also employed as a biomarker of benefit from treatment with standard chemotherapy regimens in first line NSCLC patients.

DETAILED DESCRIPTION:
VeriStrat®, a pretreatment blood-based test correlated with clinical outcome after EGFR-TKI therapy in non-small cell lung cancer (NSCLC) patients, was developed and validated in a multi-institutional study of advanced NSCLC patients treated with gefitinib [Taguchi et al] . The VeriStrat algorithm was developed using a training set of pre-treatment serum samples from patients who then experienced either long term stable disease or early progression on gefitinib therapy. Mass spectra from these patients' serum samples were used to define eight MS features (i.e. peaks), differentiating these two outcome groups. An algorithm (VeriStrat) utilizing these features and based on a k-nearest neighbors (KNN) classification scheme was created and its parameters were optimized using additional spectra from the training cohort. All aspects of VeriStrat were frozen after development. VeriStrat assigns each spectrum a "Good" or "Poor" label. VeriStrat was validated in a blinded fashion on two independent cohorts of patients who were treated with gefitinib or erlotinib. These studies confirmed that patients classified as "Good" had better outcome than patients classified as "Poor" (HR of death = 0.47 P = 0.0094 in one cohort, HR of death = 0.33 P = 0.0007 in the other).

In the original study, VeriStrat was shown to correlate with clinical outcome following EGFR-TKI therapy, but not in the chemotherapy or post-surgery setting: No statistically significant difference was seen in the overall survival of patients classified as "Good" or "Poor" from the serum from patients collected before second-line chemotherapy (HR = 0.74, 95%, P = 0.42 in one cohort (cohort B) and HR = 0.81, P = 0.54 in another (cohort C)). In a third control cohort of patients with resected early-stage NSCLC, the hazard ratio for overall survival was 0.90 (P = 0.79). However, further analysis of the subsets of chemotherapy samples demonstrated that separation between "Good" and "Poor" arms may depend on a particular type of chemotherapy. Thus a retrospective subset analysis of the cohort C showed that while patients treated with docetaxel in second line did not show any sign of separation, patients receiving a combination of platinum-based agents with either vinorelbine or gemcitabine or paclitaxel had a trend to separation between the two arms.

The working hypothesis for the mechanism is that the VeriStrat "Poor" label is related to the activation of canonical and non-canonical MAPK pathways downstream from receptor tyrosine kinases, with possible cross-talk activation of the NF-kB pathway. This means that VeriStrat may demonstrate different predictive performance depending on the particular chemotherapy treatment and its associated with cell pathway interactions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented inoperable, locally advanced (stage IIIb with supraclavicular lymph node metastases),metastatic (stage IV) or recurrent NSCLC
* Age ≥18 years
* Life expectancy more than 3 months
* ECOG performance status 0-1
* At least one unidimensionally measurable lesion (as per RECIST criteria ver 1.1)
* Adequate baseline bone marrow, hepatic and renal function
* Patients may have had prior therapy providing the following conditions are met:

Radiation therapy: wash-out period of 28 days; Surgery: wash-out period of 14 days

* Patients must give written informed consent to participate in the study

Exclusion Criteria:

* Prior chemotherapy or treatment with another systemic anti-cancer agent (for example tyrosine kinase inhibitor).
* Patients must not receive any other investigational agents while on study
* Patients with myocardial infarction within the last six (6) months, unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
* History or evidence upon physical examination of CNS disease unless adequately treated (e.g., any brain metastasis, seizure not controlled with standard medical therapy, or history of stroke).
* Patients with active or uncontrolled systemic disease/infections or with serious illness or medical conditions, which is incompatible with the protocol
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol
* Pregnancy or lactation. Patients - both males and females - with reproductive potential (i.e. menopausal for less than 1-year and not surgically sterilized) must practice effective contraceptive measures throughout the study. Women of childbearing potential must provide a negative pregnancy test (serum or urine) within 14 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by advanced non small cell lung cancer who are chemotherapy-naive and candidates for first-line chemotherapy. This population includes patients with non-squamous histology and patients with squamous histology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2011-02; Primary Completion 2017-07 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  The primary objective of this study is to evaluate the potential role of VeriStrat test as a biomarker of benefit from treatment with standard chemotherapy regimens in first line NSCLC patients in terms of progression-free survival (PFS) (primary endpoint) in two populations: patients with non-squamous histology treated with cisplatin and pemetrexed, and patients with squamous histology treated with cisplatin and gemcitabine

SECONDARY OUTCOMES:
Overall survival | 2 years
  A secondary endpoint is to evaluate the role of VeriStrat as a biomarker of the secondary endpoints overall survival, in two groups of first line patients with non-small cell lung cancer (NSCLC), described above.
Correlation with RECIST response | Every 6 weeks
  A secondary endpoint is to evaluate the possible correlation of VeriStrat classification with best RECIST responses.
Correlation with known biomarkers | Every 6 weeks
  A secondary endpoint is to evaluate the possible correlation of VeriStrat classification with the available measurements of known biomarkers: the mutation statutes of EGFR, K-RAS, and ALK, and levels of ERCC1, RRM1 and TS.
Changes of VeriStrat with disease progression | Every 6 weeks
  A secondary endpoint is to evaluate possible changes of VeriStrat classification with disease progression.
Metabolomics | Every 6 weeks
  A secondary endpoint is to identify, measure, and interpret the complex time-related concentrations, activity, and fluxes of endogenous metabolites in biosamples such as blood and urine to improve disease prognosis and monitoring; provide insight into drug metabolism and toxicology; provide a linkage between the human metabolome and the human genome and proteome.
Circulating tumor cells. | Every 6 weeks
  A secondary endpoint is isolate, identify and characterize molecularly the circulating tumor cells (CTCs) before start of treatment (within 2 weeks), at each patient's evaluation and at progression.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Grossi, MD, Principal Investigator — IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy
Locations (1):
- IRCCS Azienda Ospedaliera Universitaria San Martino - IST Istituto Nazionale per la Ricerca sul Cancro, Genoa, Italy

REFERENCES:
- [Derived] Morbelli S, Alama A, Ferrarazzo G, Coco S, Genova C, Rijavec E, Bongioanni F, Biello F, Dal Bello MG, Barletta G, Massollo M, Vanni I, Piva R, Nieri A, Bauckneht M, Sambuceti G, Grossi F. Circulating Tumor DNA Reflects Tumor Metabolism Rather Than Tumor Burden in Chemotherapy-Naive Patients with Advanced Non-Small Cell Lung Cancer: 18F-FDG PET/CT Study. J Nucl Med. 2017 Nov;58(11):1764-1769. doi: 10.2967/jnumed.117.193201. Epub 2017 Apr 27. PMID 28450567